CLINICAL TRIAL: NCT05743361
Title: Studio Sierologico in Volontari Vaccinati Contro COVID-19
Brief Title: Security Efficacy COVID-19 Vaccination
Acronym: SECVAX
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 20C121
Record Dates: First submitted 2023-02-21; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Autoimmune State; SARS-CoV-2 Infection
Keywords: SARS-CoV-2; Vaccine
MeSH Terms: conditions — Autoimmune Diseases; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autoantibodies: Detection of: ANA, AMA, anti-dsDNA, anti-ENA, anti-MPO, anti-PR3, aPL, RF, ACPA, anti- TPO, anti-TG
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Detection of ANA, AMA, anti-dsDNA, anti-ENA, anti-MPO, anti-PR3, aPL, RF, ACPA, anti- TPO, anti-TG

SUMMARY:
Preliminary data support a possible molecular mimicry between SARS-CoV-2 and autologous components. This suggests the occurrence of autoimmunity during COVID-19. Consistently, autoimmunity may occur after SARS-CoV2 vaccination. The study aims to investigate the production of autoantibodies after vaccination in healtcare workers.

DETAILED DESCRIPTION:
Healtcare workers undergoing SARS-CoV-2 vaccination (with RNA-vaccines) will be included on a voluntary basis. Blood samples will be collected before and after vaccination (1 -3 - 6 - 12 months). All the vaccination side effects will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers undergoing SARS-CoV-2 vaccination

Exclusion Criteria:

* Pregnancy
* Full blown autoimmune diseases
* Active vaccinations within 3 months before enrolment (excluding the influenza vaccine)
* Previous vaccination severe side effects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare workers undergoing SARS-CoV-2 vaccination
Sampling Method: Non-Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Autoantibody Levels | Before vaccination and 1, 6 and 12 months after vaccination
  ANA, AMA, anti-dsDNA, anti-ENA, anti-MPO, anti-PR3, aPL, RF, ACPA, anti-TPO, anti-TG

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Meroni, MD, Principal Investigator — Istituto Auxologico Italiano IRCCS
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: No